CLINICAL TRIAL: NCT05728866
Title: Effectiveness of Immersive Virtual Reality (IVR) Combined With Task-Specific Training on Hemiplegic Arm Function Following Stroke: A Single Case Series Study.
Brief Title: Effectiveness of IVR Combined With Task-Specific Training on Hemiplegic Arm Function Following Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20025720
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (VR) therapy (Experimental)
  Interventions: Procedure: VR immersive therapy

INTERVENTIONS:
Procedure: VR immersive therapy — Participants will be asked to participate in 5 consecutive, 1-hour, 1:1 therapy sessions focused on rehabilitation of their weakened arm. Each session will involve use of a Virtual Reality (VR) system to deliver an immersive environment to encourage movement of the arm. The system also relies on 6 body-worn sensors that will detect movements of participant's arms and trunk. VR use will encompass 30-minutes of the therapy session, the remainder of the session will involve working with the therapist in addressing the functional tasks that are most meaningful for the participant and that involve the upper extremities.

SUMMARY:
The purpose of this research study is to understand the efficacy of using an immersive Virtual Reality (VR) environment, with task-specific training, to encourage arm movement following stroke.

DETAILED DESCRIPTION:
The study will investigate how people who have had a stroke use their weakened arm in everyday tasks, and how this relates to measurements of movement ability from standardized clinic tests. Results of this research will ultimately help develop more effective training approaches to be used with stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Diagnosed as having an ischemic or hemorrhagic stroke (with documented confirmatory neuroimaging in the medical record) that occurred at least 6-months prior to study enrollment.
* Lack of full active range of motion in the involved shoulder, elbow, and wrist as the result of the injury.
* At the time of study enrollment, participant completed structured therapeutic interventions at least 2-months prior.
* Participants will not participate in Yoga, Tai-Chi, or other wellness lifestyle classes while participating in the study.
* Absence of significant cognitive impairment as determined by a Mini-Mental Status Examination score of greater than or equal to 24.
* The absence of upper extremity injury limiting functional use of the arm prior to the incident stroke.

Exclusion Criteria:

* Unable to provide informed consent.
* Sensory loss as determined by a score of 2 on the sensory item of the NIH Stroke Scale.
* Pain in the involved upper limb that could interfere with daily activities as evidenced by a pain score of 5 or greater on the Numeric Pain Rating Scale.
* History of greater than two strokes.
* Suffered a stroke less than 6-months prior to participating in the study.
* A history of, or being susceptible to, cyber-sickness (i.e., motion sickness).
* Unable to don/doff accelerometer independently, or the lack of support in the home to assist with donning/doffing device; and
* A history of seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in hemiplegic arm movements | Baseline to approximately 12 days
  Arm movements will be measured using wrist-worn accelerometers. Amount of movement will be measured prior to and following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Chu, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No